CLINICAL TRIAL: NCT02027415
Title: Effects of Oral Nitrate Supplementation on Vascular and Pulmonary Oxidative Stress Markers Following Traffic Pollution Exposure
Brief Title: The Effect of Juice Types on the Responses to Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Howard M. Kipen, MD, MPH, Professor and Department Chair, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2013003273
Record Dates: First submitted 2013-12-16; First posted 2014-01-06 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Air Pollution
Keywords: air pollution; food; nitrites; nitrates; breath tests/methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beet Orange (Experimental): Beet juice will be given prior to the first car ride and orange juice will be given prior to the second car ride.
  Interventions: Dietary Supplement: Beet juice; Dietary Supplement: Orange juice
- Orange Beet (Experimental): Orange juice will be given before the first car ride and beet juice will be given before the second car ride.
  Interventions: Dietary Supplement: Beet juice; Dietary Supplement: Orange juice

INTERVENTIONS:
Dietary Supplement: Beet juice — 2 cups of beet juice will be given before the car ride
Dietary Supplement: Orange juice — 2 cups of orange juice will be given before the car ride

SUMMARY:
The study hypothesis is that drinking different juices will affect the body's responses to air pollution. Subjects will be exposed to air pollution during a 2-hour car ride on the NJ (New Jersey) Turnpike. Each subject will be asked to do this twice. Before one car ride, the subject will be asked to drink orange juice. Before the other car ride, the subject will be asked to drink beet juice. Samples of blood and exhaled breath will be collected before, immediately after, and 24 hours after each car ride. Levels of nitrites/nitrates will be measured in the blood and breath.

DETAILED DESCRIPTION:
Subjects will participate in two exposure sessions. The air pollution exposure consists of a 2-hour car ride along the NJ Turnpike. Samples will be collected at 3 time points for each exposure session: pre-exposure, immediately post-exposure, and 24 hours post-exposure. Blood samples will be collected immediately before and after a 5-minute occlusion at each time point. The subject will also be asked to provide samples of exhaled breath and complete symptom and stress questionnaires at each time point.

Blood samples will be analyzed for serum nitrite. Exhaled breath samples will be analyzed for nitrates and nitrites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Must live within 20 miles of Piscataway, NJ

Exclusion Criteria:

* • Are a current smoker

  * Are pregnant or breastfeeding
  * Are HIV-positive
  * Have an active medical condition such as high blood pressure, asthma, diabetes or other serious disease
  * Have a heart condition such as atrial flutter, atrial fibrillation or a pacemaker
  * Are unable to ride comfortably in a car for 2 hours
  * Travel to the EOHSI (Environmental and Occupational Health Sciences Institute) Clinic Center on major highways for more than 3 miles (the Garden State Parkway, the New Jersey Turnpike, Routes 287, 1, 18, or 9).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in plasma nitrite concentration | Prior to the car ride, immediately after the 2-hour car ride, and 24 hours later
  Change in plasma nitrite concentration pre- and post-occlusion

SECONDARY OUTCOMES:
Change in nitrite/nitrate concentration in exhaled breath | Prior to the car ride, immediately after the 2 hour car ride and 24 hours later
  Change in nitrite/nitrate concentration in exhaled breath

CONTACTS AND LOCATIONS:
Overall Officials: Howard Kipen, MD, Principal Investigator — Rutgers RWJMS
Locations (1):
- Environmental and Occupational Health Sciences Institute, Piscataway, New Jersey, United States

REFERENCES:
- [Background] Laumbach RJ, Rich DQ, Gandhi S, Amorosa L, Schneider S, Zhang J, Ohman-Strickland P, Gong J, Lelyanov O, Kipen HM. Acute changes in heart rate variability in subjects with diabetes following a highway traffic exposure. J Occup Environ Med. 2010 Mar;52(3):324-31. doi: 10.1097/JOM.0b013e3181d241fa. PMID 20190650
- [Background] Hussain S, Laumbach R, Coleman J, Youssef H, Kelly-McNeil K, Ohman-Strickland P, Zhang J, Kipen H. Controlled exposure to diesel exhaust causes increased nitrite in exhaled breath condensate among subjects with asthma. J Occup Environ Med. 2012 Oct;54(10):1186-91. doi: 10.1097/JOM.0b013e31826bb64c. PMID 23001278
- [Background] Laumbach RJ, Kipen HM. Acute effects of motor vehicle traffic-related air pollution exposures on measures of oxidative stress in human airways. Ann N Y Acad Sci. 2010 Aug;1203:107-12. doi: 10.1111/j.1749-6632.2010.05604.x. PMID 20716291